CLINICAL TRIAL: NCT03466229
Title: Impact of Antioxidant (Androferti) Treatment on Sperm DNA Integrity
Brief Title: Impact of Antioxidant Treatment on DNA Fragmentation Index
Acronym: Androferti
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Q-Pharma (Unknown); Octean (Unknown)
Responsible Party: Principal Investigator, Aleksander Giwercman, Professor, Region Skane
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Androferti
Record Dates: First submitted 2018-03-04; First posted 2018-03-15 (Actual); Last update posted 2018-03-16 (Actual); Status verified 2018-03

CONDITIONS: Male Infertility
Keywords: sperm DNA strand breaks; antioxidants
MeSH Terms: conditions — Infertility, Male

STUDY DESIGN:
Intervention Model Description: Double blind randomised placebo controlled study
Who Masked: Investigator
Masking Description: The active compound and placebo are given a number and the list linking this number to the type of preparation (placebo or active compound) is stored by one of the sponsors (Octean)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antioxidant (Active Comparator): Androferti - 1 twice per day
  Interventions: Dietary Supplement: Androferti
- Placebo (Placebo Comparator): Placebo - 1 twice per day
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Androferti
  Arms: Antioxidant
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
Increased sperm DNA Fragmentation Index implies decreased male fertility in vivo and in vitro. There is need for developing new strategies for improvement of male fertility. The study aims to investigate whether high sperm DNA Integration Index can be treated by use of antioxidants.

DETAILED DESCRIPTION:
In the Western world, approximately 15-20% of couples experience infertility problems during their reproductive life. In this context ´'infertility' is defined as 12 months of unprotected intercourse without getting pregnant.

Although there is limited access to reliable diagnostic methods, it is assumed that in at least 50% of all cases 'male subfertility' is a contributing or the main cause of the infertility of the couple. The gold standard in assessment of male reproductive function is standard semen analysis including evaluation of sperm number, motility and morphology. Although efforts have been made in to improve and standardise the methodology for semen analysis, there are no well established cut off levels for sperm concentration, motility or morphology which accurately predict the chance of pregnancy or indicate which assisted reproductive technique (ART) - the most frequent therapy for infertility- will ultimately be the most effective. This lack of diagnostic tools is not only hampering proper management of infertility but also represents a serious limitation in relation to the understanding of biological underpinnings of the disorder and as a consequence, the development of cause related treatment modalities.

Although various novel alternative methods of assessing semen quality have been developed, so far, none have contributed to or altered our clinical approach to the treatment of infertile couples. During the passed two decades a lot of attention has been paid to impairment of sperm DNA integrity as a possible cause of male subfertility. There are different techniques currently available for the assessment of sperm DNA integrity e.g. Sperm Chromatin Structure Assay (SCSA®), Comet, TUNEL and sperm chromatin dispersion test. Generally, the use of these tests has shown an increased proportion of sperm with fragmented DNA structure among subfertile men as compared to proven fertile or men from general population. Although measuring different characteristics of the status of sperm DNA (e.g. presence of single and double strand breaks, propensity to damage and probable cause of the fragmentation), comparisons of the results obtained with two or more of these tests show a correlation coefficient of a magnitude 0.4 to 0.6, indicating that, although not completely overlapping, the tests to a certain extent assess some of the same characteristics of sperm DNA. Another interesting finding is that there is only a weak to moderate correlation between standard sperm parameters and measures of DNA integrity, the level of association (correlation coefficient ~ 0.6) the most pronounced being for motility. This means that assessment of sperm chromatin integrity adds to the information obtained by standard semen analysis.

The most appraised, standardised and studied of the sperm nDNA tests is the SCSA® which is based on a very well defined protocol for handling of samples and subsequent data analysis. The robustness of the techniques was exemplified by a comparison of the SCSA® analysis of almost 200 samples results performed by two independent laboratories which found a correlation coefficient of 0.9 with mean difference between the DNA Fragmentation Index (DFI) results of about 1%. A further advantage of the SCSA® method over the remaining assessment techniques is the relatively large number of studies that have utilised the technique in clinical settings constituting a considerable record of the method's performance in predicting fertility outcome.

Briefly, these data indicate that the chance of spontaneous pregnancy decreases at DFI levels above 20% and approaches zero if DFI exceeds 30%. This is also true for Intrauterine insemination (IUI). However, it seems that even spermatozoa from samples with high DFI can be used for in vitro fertilisation by standard IVF or ICSI, with some data suggesting that ICSI might actually be more efficient using samples with high (>30%) DFI. A finding, which may at first appear paradoxical but may be a reflection of the relative probability of fortuitously selecting a sperm with intact DNA. The data regarding fertilisation rate, embryo quality and risk of miscarriage in relation to DFI are also conflicting.

The biological mechanisms responsible for DNA strand breaks and other types of impairment of sperm DNA integrity are not completely known. Amongst others incomplete DNA repair during spermiogenesis, abortive apoptosis and/or increased level of oxidative stress have been suggested as possible options .

The overall aim of this project is to evaluate effect of restoring oxidant balance using Androferti, (Q Pharma Laboratories; Alicante, Spain) on sperm DNA integrity in subfertile men with high level of DFI.

ELIGIBILITY:
Inclusion Criteria:

1. Referred due to infertility
2. Age: 18-50 years,
3. Non-smoking,
4. Sperm DNA Fragmentation Index >25%

Exclusion Criteria:

1. Body mass index (BMI) ≥30,
2. FSH outside the normal range of 2-8 IU/L,g)
3. LH outside the normal range of 2-10 IU/L,
4. T < 10nmol/L
5. Treated with antihypertensive drugs, hormones, statins, psychotropic drugs, or oral cortisone for the last six months,
6. History of anabolic steroids use,
7. Taking antioxidant supplementation the last six months.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Men able to deliver semen sample and investigated due to infertility
Enrollment: 79 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
DFI_3 | Change in DNA Fragmentation Index from Baseline to 3 months
  3_month_change_DNA Fragmentation Index assessed by Sperm Chromatin
DFI_6 | Change in DNA Fragmentation Index from Baseline to 6 months
  6_month_change_DNA Fragmentation Index assessed by Sperm Chromatin Structure Assay

SECONDARY OUTCOMES:
Concentration_3 | Change in sperm concentration from baseline to 3 months in millions/mL
  Change sperm concentration 3 months
Concentration_6 | Change in sperm concentration from baseline to 6 months in millions/mL
  Change sperm concentration 6 months
Motility_3 | Change in sperm motility from baseline to 3 months in %
  Change sperm motility 3 months
Motility_6 | Change in sperm motility from baseline to 6 months in %
  Change sperm motility 6 months
Morphology_3 | Change in sperm morphology from baseline to 3 months in %
  Change sperm morphology 3 months
Morphology_6 | Change in sperm morphology from baseline to 6 months in %
  Change sperm morphology 6 months

IPD SHARING:
Plan to Share IPD: Undecided
Plan to share IPD has not yet been discussed

REFERENCES:
- [Derived] Stenqvist A, Oleszczuk K, Leijonhufvud I, Giwercman A. Impact of antioxidant treatment on DNA fragmentation index: a double-blind placebo-controlled randomized trial. Andrology. 2018 Nov;6(6):811-816. doi: 10.1111/andr.12547. Epub 2018 Oct 8. PMID 30298673